CLINICAL TRIAL: NCT01482364
Title: BEtter Control of Blood Pressure in Hypertensive pAtients Monitored Using the BEtter Control of Blood Pressure in Hypertensive pAtients Monitored Using the HOTMAN® sYstem
Brief Title: BEtter Control of Blood Pressure in Hypertensive pAtients Monitored Using the HOTMAN® sYstem
Acronym: BEAUTY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hemo Sapiens, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-01-2011
Record Dates: First submitted 2011-11-28; First posted 2011-11-30 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2011-11

CONDITIONS: Hypertension
Keywords: HOTMAN System; Hemodynamic integrated management
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HOTMAN-driven therapeutic approach arm (Experimental): "Hotman-driven" therapeutic approach arm(group IHM) will receive treatment according to the results of the HOTMAN® System.
  Interventions: Device: Integrated hemodynamic management (IHM) - HOTMAN System
- Control arm (Placebo Comparator): Control arm will receive usual antihypertensive care according to the 2007 ESH Guidelines.
  Interventions: Device: Non Integrated Hemodynamic Management (Non-IHM) - HOTMAN System

INTERVENTIONS:
Device: Integrated hemodynamic management (IHM) - HOTMAN System — Therapeutic approach according to HOTMAN System measurement(ICG)results .
  Arms: HOTMAN-driven therapeutic approach arm
Device: Non Integrated Hemodynamic Management (Non-IHM) - HOTMAN System — Therapeutic approach according to 2007 ESH Guidelines, regardeless HOTMAN results.
  Arms: Control arm

SUMMARY:
The purpose of this study is to demonstrate that monitoring hemodynamic parameters and then applying a predefined algorithm of drug selection (i.e. integrated hemodynamic management - IHM) improves the control of systolic blood pressure (SBP) at ambulatory blood pressure monitoring (ABPM) in hypertensive patients, as compared to classical drug selection (i.e. without IHM) during a 6 months intensive treatment program.

DETAILED DESCRIPTION:
Early BP control in hypertensives guarantees the best prevention of cardiovascular events on the long term (2007 ESH-ESC Guidelines on the Management of Hypertension; VALUE study). However, in spite of education efforts and antihypertensive drugs, blood pressure control rates remain low. The most common cause of uncontrolled BP is inadequate pharmacological treatment, because the selection of antihypertensive agents is often done independently of the hemodynamic status of the patient (volemia, peripheral resistance, cardiac inotropy, heart rate).

Several studies confirmed the value of using impedance cardiography (ICG)-derived hemodynamic data as an adjunct to therapeutic decision-making in the treatment of hypertension.

Working hypothesis: when it is possible to assess the hemodynamic status, and select accordingly the most appropriate pharmacological class of antihypertensive treatment, BP reduction occurs to a greater extent and more rapidly.

In the present study an integrated therapeutic approach (IHM-Integrated Hemodynamic Management)was applied, aiming at detecting permanent vasoconstriction and/or hypervolemia and/or hyperinotropy through the HOTMAN System, in order to select the most appropriate antihypertensive drugs.

ELIGIBILITY:
Inclusion Criteria:

* patients of either sex presenting with essential hypertension
* having sustained hypertension both at office BP (SBP>140 mmHg) and at ABPM (SBP>135 mmHg daytime)
* treated with 2 to 4 antihypertensive drugs
* aged ≥ 18 and ≤ 75 years
* after signature of the Informed Consent Form (ICF)

Exclusion Criteria:

* pregnant or lactating female
* type 1 diabetes
* patients with pacemaker (ventricular/dual chamber)
* Severe aortic insufficiency
* severe hypertension (SBP ≥ 180 mmHg and/or DBP ≥110 mmHg)
* resistant hypertension requiring at least 5 antihypertensive drugs
* secondary hypertension of any aetiology, such as renal disease, pheocromocytoma, or Cushing's syndrome
* serious disorders which may limit the ability to evaluate the efficacy or safety of the protocol, including cerebrovascular, cardiovascular, renal, respiratory, hepatic, gastrointestinal, endocrine, metabolic (criteria for metabolic syndrome), haematological, oncological, neurological, or psychiatric diseases
* history of the following pathologies within the last 6 months:
* myocardial infarction
* unstable angina pectoris
* percutaneous coronary intervention
* bypass surgery
* congestive heart failure stage III-IV
* left branch bundle block
* atrial fibrillation
* hypertensive encephalopathy
* stroke
* extreme obesity (BMI > 35)
* previously enrolled subjects
* alcohol or drug abuse in the past 2 years
* planned hospitalization during the study period
* participation in any other clinical study within 30 days prior to screening visit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2011-10; Primary Completion 2013-06 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Absolute change in daytime SBP, under ambulatory conditions (ABPM) after a 6 months follow-up. | baseline and after 6 months of treatment
  Absolute change in daytime SBP, under ambulatory conditions (ABPM) after 6 months follow-up.

SECONDARY OUTCOMES:
The percentage of normalization of SBP (<135 mmHg) at ABPM | baseline and after 6 months of treatment
  The percentage of normalization of SBP (<135 mmHg) at ABPM
The absolute change from baseline in 24h SBP-ABPM, in 24h DBP-ABPM | baseline and after 6 months of treatment
  The absolute change from baseline in 24h SBP-ABPM, in 24h DBP-ABPM
Rate of side effects | from baseline to 6 months of treatment
  Rate of side effects
The normalization of hemodynamics (CI, HR and SSVRI), the normalization of PWV and central BP | baseline and after 6 months of treatment
  The normalization of hemodynamics (CI, HR and SSVRI), the normalization of PWV and central BP

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Laurent, Principal Investigator — Hopital europeen Georges Pompidou
Locations (5):
- Tallinn Hypertension Excellence Centre, Tallinn, Estonia
- Hôpital européen Georges Pompidou, Paris, France
- Milano Hypertension Excellence Center, Milan, Italy
- University of Oslo, Ullevaal Hospital, Oslo, Norway
- Hypertension Unit, Dpt of Hypertension and diabetology, Medical University of Gdansk, Gdansk, Poland

REFERENCES:
- [Derived] Fadl Elmula FE, Rebora P, Talvik A, Salerno S, Miszkowska-Nagorna E, Liu X, Heinpalu-Kuum M, Comotti T, Larstorp AC, Rostrup M, Swierblewska E, Valsecchi MG, Kjeldsen SE, Viigimaa M, Narkiewicz K, Parati G, Laurent S; BEtter control of blood pressure in hypertensive pAtients monitored Using the HOTMAN sYstem (BEAUTY) Study Investigators. A randomized and controlled study of noninvasive hemodynamic monitoring as a guide to drug treatment of uncontrolled hypertensive patients. J Hypertens. 2015 Dec;33(12):2534-45. doi: 10.1097/HJH.0000000000000749. PMID 26485460